CLINICAL TRIAL: NCT06732414
Title: A Biorepository of Multiple Allergic Diseases (MADREP) With Longitudinal Follow-up
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001928; 001928-I
Record Dates: First submitted 2024-12-12; First posted 2024-12-13 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-26

CONDITIONS: Allergy, Sinus Disorders, Atopic Diseases, Asthma, Allergic Rhinitis, Atopic Dermatitis, EoE, Drug a
Keywords: Allergy, repository, data, sample collection
MeSH Terms: conditions — Hypersensitivity; Asthma; Rhinitis, Allergic; Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conditions that may be initially evaluated or managed by A&I but not categorized in 1 or 2 above: Conditions that may be initially evaluated or managed by an allergist-immunologist or rhinologist but not categorized in (1) or (2) above (eg, hypereosinophilia, mast cell disorders, pruritus, chronic cough, smell disorders)
- Individuals with a suspected allergic or atopic disease: Individuals with a suspected allergic or atopic disease, but without demonstrated allergen sensitization (eg, contact hypersensitivity, chronic spontaneous urticaria, drug allergy)
- Individuals with an allergic, atopic, or sinus disease: Individuals with an allergic, atopic, or sinus disease (eg, atopic dermatitis, eosinophilic esophagitis (EoE), asthma, chronic rhinosinusitis with polyposis) with documented allergen sensitization in the skin or blood

SUMMARY:
Background:

Allergic or sinus diseases can affect the skin, sinuses, airways, and other parts of the body. Examples include pollen and environmental allergies, food allergies, asthma, and eczema. To learn more about how to prevent and treat these diseases, researchers need to study data, blood, fluid, and tissue samples from people affected by them.

Objective:

To collect data, blood, fluid, and tissue samples from people with allergic or sinus diseases.

Eligibility:

People aged 3 to 100 years with allergic or sinus diseases.

Design:

Participants will have at least one clinic visit, and most participants will have a baseline visit, annual visit, and an end of study visit. The duration of the study is 1 to 3 years. During the first clinic visit, the following procedures will be done to collect data, blood, fluid, and tissue samples:

* Blood will be collected.
* Cells and fluid may be collected from the inside of the nose using a long swab, and a small piece of skin may be scraped from inside the nose.
* Skin cells will be collected by rubbing with a cotton swab.
* A urine sample will be collected.
* Allergy skin prick tests. Allergy-causing substances will be placed on the back or arm and the skin underneath gently scratched. If the participant is allergic to the substance, the skin may become red, itchy, and swollen locally ( at the site of the test).
* Lung function test. Participants will breathe into a machine that measures the air moving in and out of their lungs.
* If, as part of their routine care, participants are undergoing procedures such as having nasal polyps removed, skin tissue samples taken, or gastrointestinal biopsies, additional tissues may be collected for this study.
* Participants will complete online questionnaires regarding their symptoms, health, and life.

Participants may return for more visits for up to 3 years.

DETAILED DESCRIPTION:
Study Description:

This is a single-site repository study that will prospectively collect samples and data from participants with allergic and atopic diseases and associated conditions such as chronic rhinosinusitis and nasal polyposis, through the evaluation, testing, and monitoring of patients with these conditions at the NIH Clinical Center (CC) and via telehealth visits and/or send-in samples. This repository will provide atopic participant samples for translational studies performed by NIH investigators or their collaborators and also serve as a means for recruiting atopic control patients to ongoing NIAID and National Institute on Deafness and Other Communication Disorders (NIDCD) clinical studies.

Participants aged 3 and older will present to the NIH CC for visits for clinical evaluation and treatment of allergic diseases as appropriate. Data and samples obtained but not utilized from clinically indicated procedures will be put into the repository (e.g. physical exams, nasal endoscopy, blood tests, olfaction assessment, and nasal sinus polyp biopsy where appropriate).

Samples that may be collected prospectively for inclusion in the repository include nasal brushings, nasal lining fluid, blood, urine, and skin swabs. Additionally, extra skin, nasal sinus polyp, and gastrointestinal biopsies may be collected during clinically indicated procedures. The following assessments will also be performed for research purposes: Data collected from patient reported outcomes (PROs) and questionnaires, blood, urine, allergy skin prick testing, skin swab, and pulmonary function testing to include fractional exhaled nitric oxide testing (FeNO). Data/samples from clinical procedures will also be collected for the repository, where possible.

Although standard of care treatment may be initiated and monitored under this protocol, it will be expected that after a set number of visits outlined in the manual of operations, continued medication prescribing and monitoring will be transitioned to the referring provider, the patient s outside primary physician or allergist-immunologist, or another NIH protocol depending on the patient condition and importance for biorepository collection. No experimental treatments will be offered under this protocol.

Objective:

To create a repository of clinical, laboratory, and diagnostic data and specimens from a cohort of suspected or confirmed atopic or allergic individuals with diverse disorders seen by allergist-immunologists and rhinologists.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1)Aged 3 to 100 years.

2a) Suspected or confirmed allergic, atopic, respiratory, or nasal/sinus disorder or have suspected or confirmed history of an immune dysregulatory disorder, OR

2b) Have a clinical history of an immediate hypersensitivity reaction to aeroallergens, food, insect stings, or medications.

3) Able to provide informed consent.

4) Have or are willing to obtain a non-NIH primary physician who will manage all health conditions and be responsive for emergency medical treatment, if required.

5) Willing to allow storage of blood, skin swabs, nasal fluid/brushings, bodily fluids, and other clinically appropriate tissue specimens or data generated during participation for future use in medical research.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this

study:

1. Any condition(s) or diagnosis, physical and/or psychological, that the investigator feels precludes the patient from participation in the study.
2. For additional skin biopsies only:

   1. Individuals who have a history of keloid formation
   2. Children (<18 years old)
   3. Participants who are pregnant
3. For additional nasal-sinus polyp biopsies only:

   1. Individuals on blood thinners unless they have already been stopped for the procedure
   2. Children (<18 years old)
   3. Participants who are pregnant
4. For skin prick testing

   a. Participants who are pregnant.
5. Endoscopic Biopsy

   1. Uncontrolled asthma or Grade 3 or higher by the American Society of Anesthesiologist's Physical Status Classification System (https://www.asahq.org/standards-and-practice-parameters/statement-on-asaphysical-status-classification-system)
   2. History of adverse reaction to conscious sedation or general anesthesia required for endoscopy
   3. Hemoglobin < 11 g/dL
   4. Platelet count < 100,000 microL
   5. Pregnant or breastfeeding
   6. Severe hypoxemia due to chronic pulmonary disease
   7. Recent abdominal surgery
   8. Anticoagulant therapy that cannot be interrupted
   9. Younger than 18 years of age

Participants will be selected in an equitable manner from the available pool of potentially eligible individuals, without regard to factors such as sex, gender, race, ethnicity, sexual orientation, or socioeconomic status.

Ages: 3 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged 3 and older with suspected or diagnosed allergic diseases of varying types will be enrolled. Participants will be generally healthy, community-dwelling participants without severe medical needs requiring hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2044-11-01 (Estimated); Study Completion 2045-11-01 (Estimated)

PRIMARY OUTCOMES:
Create a repository of clinical, laboratory, and diagnostic data and specimens from a cohort of suspected or confirmed atopic or allergic individuals with diverse disorders seen by allergist-immunologists and rhinologists. | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Paneez Khoury, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD and data dictionaries will be available to researchers who request data or sample use on this protocol. IPD related to an ensuing publication for e.g. IPD related to large datasets required to be deposited will be shared with appropriate annotation by the individual researchers as required by journals and/or NIH policy, whichever is more stringent.
Supporting Information: SAP, CSR
Time Frame: As this is a biorepository it would be impossible to share all IPD in the entire study. IPD related to individual secondary use protocols will be required to be shared at the time of publication by individual investigators as well as the associated statistical analysis planned/performed. Clinical data associated with the particular study will be required to be deposited according to the DSMP
Access Criteria: IPD data sharing will occur after request/approval by the PI (or designee) and in conjunction with the procedures/approvals outlined in the appendix of the protocol. Sharing will be open to other investigators in the LAD and the NIH, and with NIDCD investigators as outlined in the associated RCA.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001928-I.html